CLINICAL TRIAL: NCT02355431
Title: A Randomized, Double-blind Phase 2 Study of Itacitinib in Combination With Erlotinib Versus Erlotinib Alone in Subjects With Stage IIIB/ IV or Recurrent Non-Small Cell Lung Cancer (NSCLC) Whose Tumors Have Epidermal Growth Factor Receptor (EGFR) Activating Mutations
Brief Title: Itacitinib in Combination With Erlotinib in Non Small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor (EGFR) Activating Mutations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn before enrolling first patient
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 39110-205
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Solid Tumors and Hematologic Malignancy; NSCLC (Non-small Cell Lung Carcinoma)
Keywords: EGFR; mutation
MeSH Terms: conditions — Hematologic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — itacitinib; INCB039110; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itacitinib plus erlotinib (Experimental)
  Interventions: Drug: Itacitinib; Drug: erlotinib
- Placebo plus erlotinib (Active Comparator)
  Interventions: Drug: erlotinib; Drug: placebo

INTERVENTIONS:
Drug: Itacitinib — tablets to be administered by mouth once daily at dose selected from safety run-in phase
  Other Names: INCB039110
  Arms: Itacitinib plus erlotinib
Drug: erlotinib — 150 mg tablets administered by mouth once daily at total daily dose of 150 mg
  Other Names: Tarceva®
Drug: placebo — matching placebo tablets to be administered by mouth at dose selected from safety run-in phase
  Arms: Placebo plus erlotinib

SUMMARY:
The purpose of this study is to determine if Itacitinib in combination with erlotinib is safe and effective in the treatment of nonsquamous non-small cell lung cancer (NSCLC) that is Stage IIIB/Stage IV or recurrent whose tumors have EGFR activating mutations.

DETAILED DESCRIPTION:
The study consists of an open-label, safety run-in to confirm the safety of Itacitinibin combination with erlotinib in subjects with nonsquamous non-small cell lung cancer (NSCLC) that is Stage IIIB, Stage IV, or recurrent whose tumors have EGFR activating mutations. Subjects in the safety run-in will receive open-label Itacitinib and erlotinib.

In the second part of the study, subjects will be enrolled and randomized to receive erlotinib (open-label) and either Itacitinib or placebo in a blinded manner. The dose of Itacitinib administered will be determined from the data produced in the safety run-in phase.

Treatment will consist of repeating 21-day cycles. Subjects will take erlotinib tablets daily and Itacitinib/placebo will be self-administered daily during the entire cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of nonsquamous NSCLC that is Stage IIIB, Stage IV, or recurrent (including Stage II).
* Documented evidence of an activating mutation in EGFR in tumor samples (exon 19 deletions or point mutation L858R in exon 21 or point mutations at codon 719).
* A mGPS of 1 or 2 as defined below:

  * Criteria: C-reactive protein >10 mg/L AND albumin ≥35 g/L Score-1
  * Criteria: C-reactive protein >10 mg L AND albumin <35 g/L Score-2
* Radiographically measurable or evaluable disease.
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate renal, hepatic, and bone marrow function demonstrated by protocol-specified laboratory parameters at the screening visit.

Exclusion Criteria:

* Known presence of the T790M mutation in EGFR in tumor samples
* Candidates for curative radiation therapy or surgery.
* Previous systemic chemotherapy for advanced disease, including EGFR inhibitor therapy, except subjects who received 1 cycle of chemotherapy while waiting to receive EGFR results, who may enroll provided that 21 days have elapsed from end of chemotherapy to the day to the baseline radiographic measurement prior to Cycle 1 Day 1.
* Distinct or suspected, or history of, pulmonary fibrosis or ILD.
* Current or previous other malignancy within 2 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive indolent or Stage I malignancy without sponsor approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Determination of the dose of itacitinib that is safe and tolerable in combination with erlotinib as measured by the number of dose-limiting toxicities (DLTs) observed in the evaluation cohort. | Baseline through Day 21
  Subjects will take erlotinib daily and begin dosing with itacitinib once daily (QD) on Cycle 1, Day 1. The safety and tolerability of the regimen will be assessed during the first 21 days of therapy
Part 2: Overall Survival (OS) | Randomization until death. Approximately 31 months.
Part 2: Progression-free survival (PFS) | Randomization to disease progression, or death due to any cause if sooner. Approximately 23 months.
  PFS is defined as the time from randomization until the earliest date of disease progression determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause if sooner.

SECONDARY OUTCOMES:
Part 2: Objective Response | Baseline through end of study. Approximately 31 months.
  Objective response determined by radiographic disease assessments per RECIST (v1.1), by investigator assessment
Part 2: Duration of Response | Baseline through end of study. Approximately 31 months.
  Duration of response determined by radiographic disease assessments per RECIST (v1.1), by investigator assessment Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Part 2: Safety and tolerability of the treatment regimens assessed by a summary of adverse events and clinical laboratory assessments. | Baseline through approximately 30 days post treatment discontinuation. Assessed after approximately 31 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard T. Kennealey, M.D., Study Director — Incyte Corporation
Locations (1):
- Ogden, Utah, United States